CLINICAL TRIAL: NCT02596425
Title: Pulmonary Recruitment Maneuver to Reduce Postlaparoscopic Shoulder Pain: Randomized Controlled Trial
Brief Title: Pulmonary Recruitment Maneuver for Postlaparoscopic Shoulder Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, Kangbuk Samsung Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-08-007
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Gynecologic Diseases
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Passive deflation (Experimental): In the controls, CO2 was removed by the traditional passive deflation of abdominal cavity.
  Interventions: Procedure: Passive deflation
- 40 cmH2O (Experimental): The intervention was five manual inflations of the lungs with positive pressure ventilation of 40 cmH2O at the end of surgery.
  Interventions: Procedure: 40 cmH2O
- 60 cmH2O (Experimental): The intervention was five manual inflations of the lungs with positive pressure ventilation of 60 cmH2O at the end of surgery.
  Interventions: Procedure: 60 cmH2O

INTERVENTIONS:
Procedure: 40 cmH2O — The intervention was five manual inflations of the lungs with positive pressure ventilation of 40 cmH2O at the end of surgery.
  Arms: 40 cmH2O
Procedure: 60 cmH2O — The intervention was five manual inflations of the lungs with positive pressure ventilation of 60 cmH2O at the end of surgery.
  Arms: 60 cmH2O
Procedure: Passive deflation — In the controls, CO2 was removed by the traditional passive deflation of abdominal cavity.
  Arms: Passive deflation

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy and safety of different recruitment maneuvers for reducing postlaparoscopic shoulder pain.

DETAILED DESCRIPTION:
Shoulder pain after laparoscopy is common and its probable mechanism is residual CO2 gas after surgery. The pulmonary recruitment maneuver can mechanically remove residual CO2 and reduce pain. In literature, there are two different recruitment maneuvers, which was manual inflation of the lungs with positive pressure ventilation of either 40cmH2O or 60cmH2O at the end of surgery. However, the higher positive pressure may be associated with more chance of barotrauma. Therefore, it is important to determine the lowest effective pressure for reducing postlaparoscopic shoulder pain. The aim of this clinical trial is to evaluate the efficacy and safety of different recruitment maneuvers (40cmH2O or 60cmH2O) for reducing postlaparoscopic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing laparoscopy for benign gynecologic diseases
* patients aged 19-65 years
* patients with american society of anesthesiology physical status I-II
* patients obtaining written informed consent

Exclusion Criteria:

* patients with chronic shoulder pain, chronic epigastric pain or chronic pain syndrome
* patients with past history of pneumothorax or any pulmonary surgical history
* patients with any shoulder surgery histories
* patients who required to conversion to open surgery from laparoscopic surgery
* patients who required to receive incidental upper abdominal surgeries due to adhesion and injury at upper abdominal cavity
* patients with inability to understand or express 10 point visual analogue scale
* intrauterine pregnant women

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Shoulder pain | after two day of procedure
  The pain score was evaluated by 10 point visual analogue scale.

SECONDARY OUTCOMES:
Wound pain | after two day of procedure
  The pain score was evaluated by 10 point visual analogue scale.

CONTACTS AND LOCATIONS:
Overall Officials: Taejong Song, MD PhD, Principal Investigator — Kangbuk Samsung Hospital
Locations (1):
- Kangbuk Samsung Hospital, Seoul, South Korea